CLINICAL TRIAL: NCT00330291
Title: Xyrem for Treatment Refractory Insomnia Due to PTSD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to inability to recruit subjects
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Thomas L. Schwartz, M.D., Assoc Professor, State University of New York - Upstate Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4975
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: PTSD; Anxiety, Post Traumatic
Keywords: PTSD; Xyrem; Sleep problems
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Parasomnias | interventions — Sodium Oxybate

INTERVENTIONS:
Drug: Xyrem

SUMMARY:
Xyrem (sodium oxybate) is an agent with the propensity to improve slow wave sleep and sleep efficiency. It is FDA approved to treat cataplexy (drop attacks) associated with narcolepsy (sleep attacks). It has been shown to be a safe and effective agent here where deep, restorative slow wave sleep improves and next day cataplexy attacks tend not to occur.

Post Traumatic Stress Disorder (PTSD) is a psychiatric illness where a patient has witnessed or been involved in a traumatic event. After the event is over, nightmares, flashbacks, avoidance of people and places associated with trauma and hyperarousal occur which is incapacitating to the patient. One major part of PTSD hyperarousal is marked insomnia with multiple awakenings at night. This resultant poor sleep is compounded by use of SSRI serotonergic antianxiety agents (ie Zoloft(sertraline)) as first line therapy which tend to degrade slow wave, restorative sleep. Patients may respond to SSRI treatment but may fail to remit as they continue to have sleep problems. PTSD patients will often fail to respond to antihistamine (Desyrel (trazodone)) and benzodiazepine GABA hypnotic agents (Restoril(temazepam)) and continue with poor, interrupted sleep. It is possible that Xyrem's ability to remarkably improve slow wave sleep may greatly help treatment refractory insomnia due to PTSD.

The author proposes an open-label study (no placebo) where 10 PTSD patients, who have failed usual PTSD treatments and have failed usual insomnia treatments in particular will be given Xyrem in addition to their current PTSD medication. The authors wish to determine if Xyrem is a safe treatment optionin this difficult-to-treat patient population.

DETAILED DESCRIPTION:
This is an open-label (no placebo) study to see if the addition of Xyrem to a subject's PTSD medication regimen will be tolerated and possibly improve insomnia. Subjects will currently be taking at least a single psychotropic agent for the treatment of PTSD, (an SSRI). Dosing will be stable for at least 4 weeks and subjects will need to report continued insomnia despite treatment. They must also have failed at least two insomnia augmentations from separate drugs classes (benzodiazepine (temezapam, zolpidem, ect.), antihistime (quetiapine, mirtazapine, trazadone, etc.), dopamine antagonist (olanzapine, quetiapine, aripiprazole, etc.) to qualify for refractory insomnia.

Subjects will complete consenting process and attend a screening visit where they will be given a MINI psychiatric diagnostic evaluation to confirm PTSD, be given a Hamilton Anxiety, a Hospital Anxiety & Depression Scale, PCL-C, Fatigue Severity Scale, Epworth Sleepiness Scale, Pittsburgh Sleep Quality Inventory, SF-12, and sleep diary evaluation to delineate current anxiety levels (secondary measure). Subjects will have to offer consent for the study team to contact their primary providers and retrieve all past and present records to show refractory history and lack of substance abuse. Subjects will undergo a brief physical exam and bloodwork and a sleep EEG will be ordered. Furthermore, a urine drug screen will be used to screen for current misuse. If subjects are taking sleeping agents, they will be appropriately washed out (tapered per cusual clinical practice and then drug free 5 times the drug's half life) prior to sleep EEG and prior to Xyrem start. In clinical practice, Xyrem use does not warrant blood monitoring, EEGs or EKGs per the FDA.

Assuming subject meets eligibility, they will start Xyrem per cataplexy dosing guidelines. Prior to titration, a 1-2 week washout of any sleeping agent will occur. Titration will then start with 2.25g at bedtime and then again 4 hours later. This drug may be flexibly increased to 4.5g (x2 doses) based upon tolerability and effectiveness. We will escalate dose if drug is toleratedbut without efficacy. Dosing will be increased if subjective sleep quantity/quality is still reported to be unchanged or if our rating scales indicate minimal to no change.

After screening visit 1 (eligibility, medical safety determination, washout, sleep EEG) subjects will return for baseline Visit 2 and start Xyrem.

They will be seen for Visit 3 after 7 days of treatment for rating scales and possible dose escalation to 6g/d.

They will be seen for Visit 4 after 14 days of treatment for rating scales and possible dose escalation to 7.5g/d.

They will be seen for Visit 5 after 21 days of treatment for rating scales and possible dose escalation to 9g/d.

They will be seen for Visit 6/termination after 28 days of treatment for rating scales, physical exam, lab work, sleep EEG.

Subjects will be called for final safety follow up one week later and 12 weeks later.

Again, liaison with the subject's provider will occur to discuss continuance of Xyrem. If provider agrees, then long term monitoring will be in the jurisdiction of this provider. If agreement is to NOT continue Xyrem, patient will be tapered or offered help in finding a clinician comfortable with the drug. There is no major issue in stopping this drug from a withdrawal point of view as it does not build up in the system over time in regards to dependence when used at bed time only. Insomnia will likely return and patient would go back to their usual treatment if desired and most likely their original level of insomnia.

Safety Measures The overall safety and tolerability of Xyrem will be assessed throughout the study by adverse event recording, clinical laboratory test results and physical exams. A Safety monitoring board will consist of the PI and two psychiatry attendings from University Hospital

ELIGIBILITY:
Inclusion Criteria:Patients are included in the study if all of the following criteria are met:

1. Written informed consent is obtained.
2. The patient is English-speaking and 18 through 64 years of age inclusive.
3. The patient meets the DSM-IV criteria for PTSD as determined by the MINI and psychiatric evaluation.
4. The patient is currently taking a medication for PTSD for ≥ 12 weeks and remains symptomatic for insomnia
5. The patient has failed to respond to at least two of the following sleeping agents (there must be at least two drug classes failed): true benzodiazepines hypnotics (temazepam), non-benzodiazepine GABA modulating hypnotics (zaleplon dosed x2 or zolpidem, an antihistamine (trazadone or mirtazapine), or an atypical antipsychotic (olanzapine or quetiapine).
6. The patient is in good health as determined by a medical and psychiatric history, medical examination, lab tests.
7. Women must be of nonchildbearing potential [i.e., postmenopausal, be surgically sterile (hysterectomy or tubal ligation)] or must meet all of the following conditions: using a reliable, medically accepted form of contraception for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; and adequate barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen). Women must be given a pregnancy test (ßHCG), unless they are at least 2 years postmenopausal or surgically sterile, and the results of the test must be negative.
8. The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

   -

Exclusion Criteria:Patients are excluded from participating in this study if 1 or more of the following criteria are met:

1. Have a primary Axis I or II psychiatric condition outside of PTSD
2. The patient is a significant risk of suicide
3. The patient has a history of substance dependence (except nicotine) ever
4. The patient has a history of substance abuse in the last 5 years
5. The patient has any serious, unresolved or unstable medical and/or psychiatric condition (treated or untreated) which makes Xyrem treatment risky. The inborn error of metabolism succinic semialdehyde dehydrogenase deficiency is contraindicated Uncontrolled hypertension, heart failure are relative contraindications due to Xyrem's high salt content
6. The patient has previously participated in any clinical study with Xyrem or treated with Xyrem.
7. The patient is a pregnant or lactating woman (women becoming pregnant during the study will be withdrawn from the study).
8. The patient has used an investigational drug within 1 month before the screening visit or is participating in a concurrent clinical trial.
9. The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery) or have an explanable medical condition causing insomnia

(k) The patient is unlikely to comply with the study protocol, be unreliable in providing ratings, or is unsuitable for any reason, as judged by the investigator.

(l) The patient has a clinically significant deviation from normal in the physical examination.

(m) The patient has a responsibility that would require them to wake up and perform within 4 hours of a Xyrem dose (n) The patient refuses to cease use of sleeping pills (o) The patient has been diagnosed with sleep apnea (we will clinically prescreen for this and check on initial EEG).

(p) If the patient lives alone, they will need to agree to being called by a member of the study team to assess the subject's well being on the morning after the first ingestion of study drug and on the morning after any dose increase to monitor for excess sedation, sleepwalking, etc. (q) If the patient lives with children less than 6 years of age, they will not be allowed in the study.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Schwartz, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States